CLINICAL TRIAL: NCT03269032
Title: Impact of the Mediterranean Diet on the Gut Microbiome and Symptoms of Diarrhea-Predominant Irritable Bowel Syndrome
Brief Title: Mediterranean Diet and the Gut Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00039422
Record Dates: First submitted 2017-08-30; First posted 2017-08-31 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2021-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: Mediterranean diet; gut microbiome; gastrointestinal
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: The study will have two phases, Phase 1 will study healthy subjects, who will follow a typical American diet for 2 weeks, and then cross-over to a Mediterranean-style diet for 2 weeks. Phase 2 will study subjects who have IBS-D. As above, they will first eat a typical American diet for 2 weeks, and then cross-over to a Mediterranean-style diet.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 Healthy Volunteers (Experimental): Healthy volunteers will eat a typical American diet for 2 weeks and then eat a Mediterranean-style diet for 2 weeks.
  Interventions: Other: American Diet; Other: Mediterranean-style Diet
- Phase 2 IBS Patients (Experimental): Participants with IBS will eat a typical American diet for 2 weeks and then eat a Mediterranean-style diet for 2 weeks
  Interventions: Other: American Diet; Other: Mediterranean-style Diet

INTERVENTIONS:
Other: American Diet — According to National Health and Nutritional Examination Survey (NHANES) data, the nutritional composition of the baseline typical American diet is 50%Carbohydrates, 15% Protein, 35% Fat, >11% Saturated Fatty Acids, <12% Monounsaturated Fatty Acids, and >8% Polyunsaturated Fatty Acids.
  Participants will receive 3 meals and 1 snack for each day during the study period.
Other: Mediterranean-style Diet — The nutritional composition of the baseline typical Mediterranean-style diet is 46% Carbohydrates/Alcohol (red wine will be included in the Mediterranean diet only), 17% Protein, 32% Fat, <7% Saturated Fatty Acids, >18% Monounsaturated Fatty Acids and <5% Polyunsaturated Fatty Acids.
  Participants will receive 3 meals and 1 snack for each day during the study period.

SUMMARY:
This study will evaluate the impact of a Mediterranean-style diet on microbiome diversity compared to a typical American diet. The study will observe the microbiome composition comparisons in healthy volunteers as well as in patients with Irritable Bowel Syndrome with Diarrhea (IBS-D) to see if the consumption of a Mediterranean-style diet has a positive effect on improving symptoms of IBS-D.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is the most prevalent and well-studied functional gastrointestinal disorder. While IBS has no direct mortality, it does compromise quality of life, incurs morbidity, and has a substantial economic impact on society. The gut microbiome may play a significant role in the pathogenesis of IBS. Even though the exact mechanisms underlying this relationship have not been presented, it is suggested that certain microorganisms may increase gut permeability, activate the mucosal immune response, increase visceral sensitivity and alter intestinal motility via a bidirectional brain-gut interaction. Recent studies suggest that the salutary impact of the Mediterranean diet may be due to its effects on the composition of the gut microbiome. In a recent cohort study in Italy, subjects who adhered most closely to a classical Mediterranean diet had more favorable bacterial enterotypes (e.g., Prevotella) in their stool, as well as higher levels of short-chain fatty acids - which are essential for colonic function. Studies have also showed that diet alters the predominant microbiome enterotypes and that microbiome composition can change quickly, within 24 hours, after a dietary intervention. Therefore, consumption of a Mediterranean diet may ameliorate the gut dysbiosis associated with IBS-D.

ELIGIBILITY:
Inclusion Criteria:

* must be willing to eat pre-prepared foods for 4 weeks
* subjects must have no medical, religious, or cultural dietary restrictions that would preclude their eating a Mediterranean diet.
* Phase 2 subjects- must have diagnosis of IBS based on Rome III criteria and have diarrhea-predominant disease, defined as >50% of bowel movements characterized as diarrhea

Exclusion Criteria:

* history of gastrointestinal disease, including celiac disease, inflammatory bowel disease, or lactose intolerance
* diabetes mellitus
* congestive heart failure
* coronary artery disease
* chronic liver disease or end stage renal disease
* pregnancy or breastfeeding
* trainees under the direct supervision of the PI and patients receiving direct ongoing medical care from the PI or Co-I will not be enrolled as subjects in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Phase 1- Change in predominant enterotypes and diversity of fecal microbiota | Baseline, 2 weeks, 4 weeks
  Fecal microbiota diversity and enterotypes will be determined through bacterial 16S rRNA gene sequences on stool samples collected from the healthy volunteer participants in phase 1.The data will initially be analyzed by calculating descriptive statistics and plotting to examine for potential outliers and the necessity for data transformation.
Phase 2-Change in predominant enterotypes and diversity of fecal microbiota | Baseline, 2 weeks, 4 weeks
  Fecal microbiota diversity and enterotypes will be determined through bacterial 16S rRNA gene sequences on stool samples and rectal biopsies performed on the subjects with IBS-D in phase 2.The data will initially be analyzed by calculating descriptive statistics and plotting to examine for potential outliers and the necessity for data transformation.

SECONDARY OUTCOMES:
Changes in plasma inflammatory marker - Erythrocyte sedimentation rate (ESR) | Baseline, 2 weeks, 4 weeks
  A plasma inflammatory marker that will be analyzed is the Erythrocyte sedimentation rate (ESR). Data will be analyzed in comparison of time points Baseline, 2 weeks and 4 weeks.
Changes in plasma inflammatory marker - C-reactive protein (CPR) | Baseline, 2 weeks, 4 weeks
  A plasma inflammatory marker that will be analyzed is C-reactive protein (CRP). The CRP is measured through a blood test. A CRP level of 10mg/L or lower is considered to be normal. A higher CRP indicates that their is inflammation in the body.Data will be analyzed in comparison of time points Baseline, 2 weeks and 4 weeks.
Changes in IBS Symptom Severity Scores | Baseline, 2 weeks, 4 weeks
  The IBS Severity Scoring System is a validated measure to assess the severity of IBS symptoms, and can help monitor response to treatment. Each of the 5 questions generates a score from 0-100 points with a maximum total score of 500 points. Mild IBS=75-174 points, moderate IBS=175-299 points, and severe IBS=300 points of more.Data will be analyzed in comparison of time points Baseline, 2 weeks and 4 weeks.
Changes in Hospital Anxiety and Depression Scores | Baseline, 2 weeks, 4 weeks
  Hospital Anxiety and Depression Scores (HADS) is a self assessment scale designed to detect states of depression, anxiety, and emotional distress in patients who are being treated for a clinical problem. The scale has 14 questions that are scored on a scale of 0-3, with 3 indicating higher symptom frequencies. Scores for each subscale (anxiety and depression) range from 0 to 21 with scores categorized as follows: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21. Scores for the entire scale (emotional distress) range from 0 to 42, with higher scores indicating more distress.Data will be analyzed in comparison of time points Baseline, 2 weeks and 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Weinberg, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Heath, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cresci GA, Bawden E. Gut Microbiome: What We Do and Don't Know. Nutr Clin Pract. 2015 Dec;30(6):734-46. doi: 10.1177/0884533615609899. Epub 2015 Oct 8. PMID 26449893
- [Background] Canavan C, West J, Card T. Review article: the economic impact of the irritable bowel syndrome. Aliment Pharmacol Ther. 2014 Nov;40(9):1023-34. doi: 10.1111/apt.12938. Epub 2014 Sep 9. PMID 25199904
- [Background] Shanahan F, Quigley EM. Manipulation of the microbiota for treatment of IBS and IBD-challenges and controversies. Gastroenterology. 2014 May;146(6):1554-63. doi: 10.1053/j.gastro.2014.01.050. Epub 2014 Jan 28. PMID 24486051
- [Background] Del Chierico F, Vernocchi P, Dallapiccola B, Putignani L. Mediterranean diet and health: food effects on gut microbiota and disease control. Int J Mol Sci. 2014 Jul 1;15(7):11678-99. doi: 10.3390/ijms150711678. PMID 24987952
- [Background] De Filippis F, Pellegrini N, Vannini L, Jeffery IB, La Storia A, Laghi L, Serrazanetti DI, Di Cagno R, Ferrocino I, Lazzi C, Turroni S, Cocolin L, Brigidi P, Neviani E, Gobbetti M, O'Toole PW, Ercolini D. High-level adherence to a Mediterranean diet beneficially impacts the gut microbiota and associated metabolome. Gut. 2016 Nov;65(11):1812-1821. doi: 10.1136/gutjnl-2015-309957. Epub 2015 Sep 28. PMID 26416813
- [Background] Mayer EA, Savidge T, Shulman RJ. Brain-gut microbiome interactions and functional bowel disorders. Gastroenterology. 2014 May;146(6):1500-12. doi: 10.1053/j.gastro.2014.02.037. Epub 2014 Feb 28. PMID 24583088
- [Background] De Filippo C, Cavalieri D, Di Paola M, Ramazzotti M, Poullet JB, Massart S, Collini S, Pieraccini G, Lionetti P. Impact of diet in shaping gut microbiota revealed by a comparative study in children from Europe and rural Africa. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14691-6. doi: 10.1073/pnas.1005963107. Epub 2010 Aug 2. PMID 20679230
- [Background] Wu GD, Chen J, Hoffmann C, Bittinger K, Chen YY, Keilbaugh SA, Bewtra M, Knights D, Walters WA, Knight R, Sinha R, Gilroy E, Gupta K, Baldassano R, Nessel L, Li H, Bushman FD, Lewis JD. Linking long-term dietary patterns with gut microbial enterotypes. Science. 2011 Oct 7;334(6052):105-8. doi: 10.1126/science.1208344. Epub 2011 Sep 1. PMID 21885731
- [Background] Wang Q, Garrity GM, Tiedje JM, Cole JR. Naive Bayesian classifier for rapid assignment of rRNA sequences into the new bacterial taxonomy. Appl Environ Microbiol. 2007 Aug;73(16):5261-7. doi: 10.1128/AEM.00062-07. Epub 2007 Jun 22. PMID 17586664
- [Background] Schloss PD, Westcott SL, Ryabin T, Hall JR, Hartmann M, Hollister EB, Lesniewski RA, Oakley BB, Parks DH, Robinson CJ, Sahl JW, Stres B, Thallinger GG, Van Horn DJ, Weber CF. Introducing mothur: open-source, platform-independent, community-supported software for describing and comparing microbial communities. Appl Environ Microbiol. 2009 Dec;75(23):7537-41. doi: 10.1128/AEM.01541-09. Epub 2009 Oct 2. PMID 19801464
- [Background] Weinberg RB, Dantzker C, Patton CS. Sensitivity of serum apolipoprotein A-IV levels to changes in dietary fat content. Gastroenterology. 1990 Jan;98(1):17-24. doi: 10.1016/0016-5085(90)91285-e. PMID 2104541
- [Background] McCombs RJ, Marcadis DE, Ellis J, Weinberg RB. Attenuated hypercholesterolemic response to a high-cholesterol diet in subjects heterozygous for the apolipoprotein A-IV-2 allele. N Engl J Med. 1994 Sep 15;331(11):706-10. doi: 10.1056/NEJM199409153311104. PMID 8058077
- [Derived] Mishra SP, Wang B, Jain S, Ding J, Rejeski J, Furdui CM, Kitzman DW, Taraphder S, Brechot C, Kumar A, Yadav H. A mechanism by which gut microbiota elevates permeability and inflammation in obese/diabetic mice and human gut. Gut. 2023 Oct;72(10):1848-1865. doi: 10.1136/gutjnl-2022-327365. Epub 2023 Mar 22. PMID 36948576

DOCUMENTS (1):
  • Informed Consent Form (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/32/NCT03269032/ICF_000.pdf